CLINICAL TRIAL: NCT03373240
Title: Targeting Self-regulatory Deficits Through Cognitive Remediation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000021496; 2P50DA009241-21 (NIH)
Record Dates: First submitted 2017-12-08; First posted 2017-12-14 (Actual); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Drug Use Disorders
Keywords: Drug use Disorders; Cognitive Remediation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either a (1) cognitive remediation program (training tasks) specifically designed to address cognitive-affective dysregulation or (2) control tasks (verbal fluency tasks).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU plus Cognitive Remediation Program (Experimental): Treatment normally received at this clinic that generally includes individual or group sessions and regular urine monitoring PLUS computerized games that focus on learning and decision making.
  Interventions: Behavioral: TAU plus Cognitive Remediation Program
- TAU plus Control Tasks (Placebo Comparator): Treatment normally received at this clinic that generally includes individual or group sessions and regular urine monitoring PLUS a series of computerized word games.
  Interventions: Behavioral: TAU plus Control Tasks

INTERVENTIONS:
Behavioral: TAU plus Cognitive Remediation Program — Treatment normally received at this clinic that generally includes individual or group sessions and regular urine monitoring PLUS computerized games that focus on cognitive-affective self-regulatory processes.
  Arms: TAU plus Cognitive Remediation Program
Behavioral: TAU plus Control Tasks — Treatment normally received at this clinic that generally includes individual or group sessions and regular urine monitoring PLUS a series of computerized word games.
  Arms: TAU plus Control Tasks

SUMMARY:
We are proposing a small randomized clinical trial in which 100 substance users will complete the existing Psychotherapy Development Center (PDC) pretreatment assessment battery as well as a novel battery of assays to evaluate cognitive-affective functioning. After completing pretreatment assessments, participants will be randomized to either a (1) cognitive remediation program (training tasks) specifically designed to address cognitive-affective dysregulation or (2) control tasks (verbal fluency tasks). Tasks will be completed twice per week for 4 weeks, after which assessment batteries will be repeated. Finally, we will evaluate real-world behavior and the durability of the training via a one-month follow-up, which will include assessment of substance use as well as the cognitive-affective battery.

DETAILED DESCRIPTION:
Participants will be 100 individuals (aged 18 to 50) enrolled in outpatient (non- methadone/buprenorphine) treatment for any substance use disorder (other than PCP) at the Substance Abuse Treatment Unit in New Haven. As the goal of this project is to develop interventions that address self-regulation across multiple disorders, we will recruit individuals who have a range of substance use disorders and levels of severity. Our primary Specific Aim will be to evaluate the efficacy of the cognitive-remediation program relative to the control condition control on the indicators of cognitive-affective functioning and substance use, testing the hypothesis that individuals randomized to the cognitive remediation program will demonstrate improved functioning on the cognitive-affective battery as well as reduced real-world substance abuse. We will also explore potential moderators of response to the training, including baseline measures of cognitive-affective function.

ELIGIBILITY:
Inclusion Criteria:

* Meet current DSM-5 criteria for an alcohol, stimulant, cannabis, or opioid use disorder.
* Are sufficiently stable for 4 weeks of outpatient treatment.
* Are willing to provide locator information.
* Are fluent in English and have a 4th grader or higher reading level

Exclusion Criteria:

* Meet DSM-5 criteria for a bipolar or schizophrenic disorder.
* Who have a legal case pending such that incarceration during the 4-week protocol is likely.
* Are physically dependent on alcohol, opioids or benzodiazepines or who report recent PCP use.
* Have a baseline Shipley estimated IQ less than 70
* Have 3 or more head injuries with loss of consciousness for over 30 minutes or lasting effects
* Have a history of chronic illness or neurological disorders (e.g., epilepsy or stroke) that would complicate evaluation of effects of cognitive training

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Baskin-Sommers, PhD, Principal Investigator — Yale University
Locations (1):
- Substance Abuse Treatment Center (SATU), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAU Plus Cognitive Remediation Program | TAU Plus Control Tasks
Started | 22 | 24
4-week Post Treatment | 14 | 23
Completed | 11 (This is the 1-month post follow-up) | 20 (This is the 1-month post follow-up)
Not Completed | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAU Plus Cognitive Remediation Program | TAU Plus Control Tasks | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 24 | 46
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (8.1) | 32.4 (8.6) | 33.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 15 | 19 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 12 | 17 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change in Stop Signal Reaction Time
Description: Improved functioning on cognitive-affective battery: Examining Stop Signal reaction time changed across the 4-week training period. A change score was calculated. A negative number indicates better inhibition over time.
Time Frame: Training visit 1 through 4 weeks of training
Population: All participants who completed one or more sessions of the computerized Stop Signal task. Negative change reflects improved inhibition over time.
Measure: Mean (Standard Error); unit: ms
Arm/Group | TAU Plus Cognitive Remediation Program | TAU Plus Control Tasks
Number analyzed (Participants) | 21 | 0
ms | -8.62 (2.79) |
Statistical Analysis 1: Comparison: TAU Plus Cognitive Remediation Program; Test type: Other — Examining stop signal reaction time changed across the 4-week training period; p = .003, Mixed Models Analysis; Mean Difference (Net) = -8.62, 95% CI 2-sided [-14.17 to -3.06], Standard Error of Mean 2.79

2. Primary Outcome: Change From Pre-Post in Substance Use
Description: The cube root of the number of days the participant endorsed using their primary substance. The number of days was submitted to a cube root transformation given skewness and a change score was calculated (post minus pre). A negative number indicated decreased substance use over time.
Time Frame: 4 weeks before First Training Session through the 4-week training period
Population: All participants who completed the pre- and post-treatment substance use calendar.
Measure: Mean (Standard Error); unit: cube root (number of days)
Arm/Group | TAU Plus Cognitive Remediation Program | TAU Plus Control Tasks
Number analyzed (Participants) | 15 | 19
cube root (number of days) | -.34 (.19) | .19 (.17)
Statistical Analysis 1: Comparison: TAU Plus Cognitive Remediation Program vs TAU Plus Control Tasks; Test type: Superiority; p = .049, ANOVA; Mean Difference (Net) = -.075, 95% CI 2-sided [-.333 to .184], Standard Error of Mean .127

3. Primary Outcome: Change in Pre-Post Cognitive Affective Battery- Negative Urgency Subscale (Part of the Urgency, Premeditation (Lack of), Perseverance (Lack of), Sensation Seeking, Positive Urgency, Impulsive Behavior Scale)
Description: Negative urgency (NU) subscale. The scale score range is 11-44. Higher values indicate stronger agreement with this pathway toward impulsivity. A change score was calculated. A negative number indicates less agreement with negative urgency.
Time Frame: from the week prior to training to the week after training
Population: All participants who completed the UPPS-NU for both pre- and post-treatment cognitive-affective battery
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | TAU Plus Cognitive Remediation Program | TAU Plus Control Tasks
Number analyzed (Participants) | 15 | 23
score on scale | -3.13 (1.57) | -.70 (1.27)
Statistical Analysis 1: Comparison: TAU Plus Cognitive Remediation Program vs TAU Plus Control Tasks; Test type: Superiority; p = .236, ANOVA; Mean Difference (Net) = -1.914, 95% CI 2-sided [-3.965 to .136], Standard Error of Mean 1.011

4. Primary Outcome: Change in Experimental Performance-Change in Percentage of Risky Choices Under Risk Condition of the Lottery Task
Description: The percent of risky choices per session. This would indicate that the participant selected the lottery option that reflected a riskier bet.
  A change score was calculated. A negative number indicates improved decision-making (selecting fewer risky options).
Time Frame: Training visit 1 through 4 weeks of training
Population: All participants who completed one or more sessions of the Lottery Task. Negative change indicated improved decision-making
Measure: Mean (Standard Error); unit: percent of risky choices
Arm/Group | TAU Plus Cognitive Remediation Program | TAU Plus Control Tasks
Number analyzed (Participants) | 20 | 0
percent of risky choices | -1.62 (0.77) |
Statistical Analysis 1: Comparison: TAU Plus Cognitive Remediation Program; Test type: Other — Examining whether percentage of risky choices decreased across the 4-wwek training period; p = .039, Mixed Models Analysis; Mean Difference (Net) = -1.62, 95% CI 2-sided [-3.15 to -.08], Standard Error of Mean .77

5. Primary Outcome: Change in Experimental Performance- Change in Percentage of Ambiguous Choices Under 24% Ambiguity in Lottery Task
Description: Percent of choices the participant made that reflected selecting the ambiguous option.
  A change score was calculated. A negative number reflects improved decision-making (selecting more safe options).
Time Frame: Training visit 1 through 4 weeks of training
Population: All participants who completed one or more sessions of the computerized Lottery task. Negative change reflects improved decision-making.
Measure: Mean (Standard Error); unit: percent of ambiguous choices
Arm/Group | TAU Plus Cognitive Remediation Program | TAU Plus Control Tasks
Number analyzed (Participants) | 20 | 0
percent of ambiguous choices | -1.77 (.82) |
Statistical Analysis 1: Comparison: TAU Plus Cognitive Remediation Program; Test type: Other; p = .035, Mixed Models Analysis; Mean Difference (Net) = -1.77, 95% CI 2-sided [-3.40 to -.13], Standard Error of Mean .82

6. Primary Outcome: Change in Experimental Performance- Paced Auditory Serial Addition Test (PASAT)
Description: Estimated change in percentage of trial attempts on round 3 of the PASAT. A positive number reflects more trial attempts in the third round of PASAT.
Time Frame: from the week prior to training (pre) to the week after training (post)
Population: All participants who completed one or more sessions of the computerized PASAT. Positive change reflects improved cognitive-affective functioning (distress tolerance) over time.
Measure: Mean (Standard Error); unit: percentage of trials attempted
Arm/Group | TAU Plus Cognitive Remediation Program | TAU Plus Control Tasks
Number analyzed (Participants) | 21 | 0
percentage of trials attempted | 4.26 (.57) |
Statistical Analysis 1: Comparison: TAU Plus Cognitive Remediation Program; Test type: Other; p < .001, Mixed Models Analysis; Mean Difference (Net) = 4.26, 95% CI 2-sided [3.12 to 5.39], Standard Error of Mean .57

7. Primary Outcome: Change in Pre-Post Cognitive Affective Battery: Digit Backwards
Description: Score on digit backwards. Fourteen strings of varying lengths (2 to 7 digits) are presented. A participant receives a point for each string they correctly repeat backwards. Range 0-14 points. Change score was calculated-positive values indicate improved working memory over time.
Time Frame: from the week prior to training (pre) to the week after training (post)
Population: All participants who completed the digit backwards for both pre- and post-treatment cognitive-affective battery
Measure: Mean (Standard Error); unit: scores on scale
Arm/Group | TAU Plus Cognitive Remediation Program | TAU Plus Control Tasks
Number analyzed (Participants) | 13 | 19
scores on scale | 2.08 (.62) | -.21 (.51)
Statistical Analysis 1: Comparison: TAU Plus Cognitive Remediation Program vs TAU Plus Control Tasks; Test type: Superiority; p = .008, ANOVA; Mean Difference (Net) = .933, 95% CI 2-sided [.111 to 1.755], Standard Error of Mean .403

8. Primary Outcome: Change in Pre-Post Cognitive Affective Battery: Breath Holding
Description: Negative emotionality-distress tolerance as measured by the difference between when the participant says they are uncomfortable and when they let go of holding their breath. Measured in seconds (this was natural log-transformed due to skewness for analyses). Positive change indicates improved distress tolerance over time.
Time Frame: from the week prior to training (pre) to the week after training (post)
Population: All participants who completed the breath holding task for both pre- and post-treatment cognitive-affective battery
Measure: Mean (Standard Error); unit: ln(seconds)
Arm/Group | TAU Plus Cognitive Remediation Program | TAU Plus Control Tasks
Number analyzed (Participants) | 15 | 23
ln(seconds) | .19 (.15) | -.16 (.12)
Statistical Analysis 1: Comparison: TAU Plus Cognitive Remediation Program vs TAU Plus Control Tasks; Test type: Superiority; p = .077, ANOVA; Mean Difference (Net) = .019, 97% CI 2-sided [-.177 to .214], Standard Error of Mean .096

9. Primary Outcome: Change in Pre-Post Cognitive Affective Battery: Perceived Stress Scale
Description: Negative emotionality-perceived stress. The total score ranges from 0-4. Higher scores indicate a higher level of perceived stress. A change score was calculated. Negative change indicates an improvement (reduction in perceived stress) over time.
Time Frame: from the week prior to training (pre) to the week after training (post)
Population: All participants who completed the perceived stress scale (PSS) for both pre- and post-treatment cognitive-affective battery
Measure: Mean (Standard Error); unit: scores on scale
Arm/Group | TAU Plus Cognitive Remediation Program | TAU Plus Control Tasks
Number analyzed (Participants) | 15 | 23
scores on scale | -.53 (1.38) | -1.61 (1.11)
Statistical Analysis 1: Comparison: TAU Plus Cognitive Remediation Program vs TAU Plus Control Tasks; Test type: Superiority; p = .547, ANOVA; Mean Difference (Net) = -.964, 95% CI 2-sided [-4.822 to 2.895], Standard Error of Mean 1.902

10. Primary Outcome: Change in Pre-Post Cognitive Affective Battery: Delay Discounting
Description: Incentive salience- delay discounting. Five-Trial Adjusting-Delay Discounting Task (Koffarnus & Bickel, 2014) is a 5-item behavioral assessment used to estimate the extent to which individuals prefer smaller immediate rewards over larger delayed rewards. A discount rate (ln (k)) is calculated for each time the measure is used. Discount rates for the 5- trial delay task were calculated by taking the inverse of the obtained Effective Delay 50 value, which is equivalent to the value of k, when fitted to this singular point. Ln(k) is the natural log of the discount rate. A change score was calculated. Negative change indicates improved decision-making
Time Frame: from the week prior to training (pre) to the week after training (post)
Population: All participants who completed the delay discounting task for both pre- and post-treatment cognitive-affective battery
Measure: Mean (Standard Error); unit: ln(k)
Arm/Group | TAU Plus Cognitive Remediation Program | TAU Plus Control Tasks
Number analyzed (Participants) | 15 | 23
ln(k) | -.23 (.52) | -.76 (.42)
Statistical Analysis 1: Comparison: TAU Plus Cognitive Remediation Program vs TAU Plus Control Tasks; Test type: Superiority; p = .436, ANOVA; Mean Difference (Net) = -.532, 95% CI 2-sided [-1.805 to .742], Standard Error of Mean .628

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | TAU Plus Cognitive Remediation Program | TAU Plus Control Tasks
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/22 | 1/24
Other Adverse Events (participants affected / at risk) | 0/22 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAU Plus Cognitive Remediation Program (N=22) | TAU Plus Control Tasks (N=24)
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1)
Hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hospitalization (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT03373240/SAP_003.pdf
  • Informed Consent Form (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT03373240/ICF_004.pdf
  • Study Protocol (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT03373240/Prot_005.pdf